CLINICAL TRIAL: NCT05629013
Title: TEAMS R34 #1 After-Action Reviews in Child Welfare Services
Acronym: R34-1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Danielle Fettes, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 803821; P50MH126231-01A1 (NIH)
Record Dates: First submitted 2022-11-02; First posted 2022-11-29 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Mental Health Issue; Children, Adult
Keywords: Child Welfare Services; Team Effectiveness Research; Shared Decision Making

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Child Family Team (CFT) as Usual (No Intervention): The CFT is a family meeting model that is an existing mechanism being implemented systemwide in San Diego County Child Welfare Services (CWS). Each child or youth is required to have a CFT meeting within sixty days of entering the CWS to identify areas of behavioral, emotional, or social needs, and to complete an initial case Action Plan.
- Child Family Team (CFT) with After Action Review (AAR) (Experimental): CFT is being augmented with the after-action review.
  Interventions: Behavioral: After-Action Review

INTERVENTIONS:
Behavioral: After-Action Review — After-action reviews, or debriefs, are a relatively simple, inexpensive, and quick, tool to improve learning, performance, and the effectiveness of teams and individuals. After-action reviews are active self-learning processes wherein participants reflect on specific performance episode to actively engage in self-discovery and improve learning in a non-punitive/non-judgmental manner to result in enhanced performance. This proposal aims to apply the team effectiveness intervention of the after-action review (AAR) to the services intervention of the Child and Family Team (CFT) meetings currently used in the CWS.
  Arms: Child Family Team (CFT) with After Action Review (AAR)

SUMMARY:
This project proposes to improve successful mental health service linkage in Child Welfare Services (CWS) by adapting and testing the After Action Review (AAR) team effectiveness intervention to augment the Child Family Team (CFT) services intervention. Despite being both required and a collaborative approach to service planning, CFT meetings are implemented with questionable fidelity and consistency, rarely including children and families as intended. By inclusion of child and family voice, the AAR-enhanced CFT should lead to increased fidelity to the CFT intervention and greater levels of parental satisfaction with the service and shared decision-making, thus resulting in enhanced follow-through with Action Plans and linkage to mental health care for children.

DETAILED DESCRIPTION:
The proposed project will address the following aims:

Aim 1. Conduct a qualitative needs assessment targeting the ongoing implementation of the CFT services intervention in a large, publicly funded, CWS. A qualitative inquiry consisting of interviews and focus groups with key stakeholders will result in the preparation of an action plan to address identified gaps between the current and desired CFT services intervention outcomes.

Aim 2. Adapt and tailor the AAR implementation strategy to address the CFT services intervention needs.

Aim 3. Assess mechanisms of the AAR team effectiveness intervention for CFT implementation.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for CWS leaders and/or caseworkers

1. (For leaders) Employed as one of several CWS leadership positions: CWS Director, CWS Deputy Director, CWS Regional Manager; (For caseworkers) Employed as a caseworker in one of the two participating regions for the proposed study.
2. Plans to remain employed for at least six months beyond study initiation
3. Speaks English or Spanish

Inclusion Criteria for formal and informal CFT members

1. Member of CFT with one of the participating CWS caseworkers. CFT members can include mental health services provider, Court Appointed Special Advocate (CASA), educational representative, and other supports
2. Speaks English or Spanish

Inclusion Criteria for parents/caregivers with active CWS cases

1. Parent/caregiver of child aged 6-17 with an open CWS case
2. Initial CFT meeting for open CWS case has not yet been held (Aim 3)
3. Speaks English or Spanish

Inclusion Criteria for children with active CWS cases (for mental health service linkage data extraction only*)

1. Child aged 6-17 with an open CWS case
2. Mental health services need/s (identified by the CWS caseworker via CANS screening in advance of the initial CFT meeting, during which consensus is reached regarding the Action Plan and service referral)

Exclusion Criteria:

Individuals who do not meet inclusion criteria are not eligible to participate in this study.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2023-07-28 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Collaboration & Satisfaction About Care Decisions (CSACD) | through study completion, ~9 months
  The 6-item collaboration subscale assesses collaboration, shared responsibilities for planning, open communication, and coordination. The 3-item satisfaction subscale assesses satisfaction with the decision-making process, and satisfaction with the decision itself. Although originally developed about care decisions for intensive care patients, it has since been used to measure collaboration and satisfaction with treatment planning plans associated with after-action reviews. Each participant will complete the CSACD immediately following their completion of the intervention (<1 hour). Participants respond on a 7-point likert-type scale ranging from 1=strongly disagree to 7=strongly agree. Subscale scores are computed by calculating the average item response for items representing collaboration, and items representing satisfaction, respectively. Only including the subscales regarding satisfaction.
San Diego (SD) County Behavioral Health Administrative Data | through study completion, ~9 months
  During the CFT meetings, behavioral health needs initially screened via the CANS assessment will likely be confirmed for many child/families with open CWS cases. For children/families with behavioral health treatment plans, SD County Behavioral Health Administrative Data will be assessed to determine successful service linkage.
Mathieu Team Processes Scale | through study completion, ~9 months
  The 10 first-order constructs (e.g. strategy formulation, coordination, conflict management) map to three second order constructs (i.e. transition, action, and interpersonal). This measure will be administered to CFT+AAR participants immediately following completion of the CFT+AAR intervention (<1 hour) to assess the team process of the CFT. Participants respond on a scale ranging from 1=Not at all to 5=to a very great extent, and scale scores are computed by calculating the average item response. Participants respond to questions regarding goal specification, strategy formulation, and coordination.

SECONDARY OUTCOMES:
Acceptability, Feasibility, and Appropriateness of Intervention Measure | through study completion, ~9 months
  This 9-item measure will be administered to CFT+AAR participants immediately following completion of the CFT+AAR intervention (<1 hour) to assess the extent to which the After-Action Review is appealing, liked, and welcomed in their setting (acceptability); fitting, suitable, and applicable in their setting (appropriateness); possible and doable in their setting (feasible). Each of the 9 items is rated using the following response options: 1=completely disagree, 2=disagree, 3=neither agree nor disagree, 4=agree, and 5=completely agree. Three subscales can be created by averaging responses for items representing acceptability, appropriateness, and feasibility, respectively.
Participant demographics professional characteristics | through study completion, ~9 months
  Participant age, gender, race, ethnicity, marital status, education level, primary language, and working status/profession will be collected of all participants immediately following completion of the intervention (<1 hour).
Card-Sorting Task | through study completion, ~9 months
  Card sorting elicits individual mental models to understand how participants structure their knowledge. In open card sorts participants are provided with a set of key concepts and asked to sort them into categories. Each participant then creates a label for each category. In closed card sorts, participants are similarly given a set of key concepts, but participants are given pre-defined categories that each concept must be sorted into. Within team environments, card sorting can be used to examine the degree to which team members are thinking about key concepts in a similar manner (e.g., team mental models) by comparing the categories and sorted content across members. For this proposal, each participant will complete the card sorting task immediately following completion of the intervention (<1 hour). In doing so, the concepts contained in the card sort will be representative of specific CFT roles, task responsibilities, and goals.
McAllister Affect-Based Trust | through study completion, ~9 months
  This 5-item scale assesses perceptions of affect-based trust amongst CFT members. Items center on individual's perceptions that team members can share ideas freely, that team members listen to one another, that team members care for one another, and that team members are invested in working well with one another. Each participant will complete the WAI-SR immediately following their completion of the intervention (<1 hour). Participants respond on a scale ranging from 1=strongly disagree to 7=strongly agree, and scale scores are computed by calculating the average item response.
Psychological Safety | through study completion, ~9 months
  Edmondson's 7-item Psychological Safety Climate Measure evaluates perceptions of the work environment (in this case, the CFT meeting) as being one wherein policies and procedures foster a safe and comfortable space for interpersonal risk. Each participant will complete the Psychological Safety Climate Measure immediately following their completion of the intervention (<1 hour). Participants respond on a scale ranging from 0=doesn't apply at all to 4=entirely applies, and overall scale scores are computed by calculating the average item response.
State-Wide CFT Fidelity Tool | through study completion, ~9 months
  The CFT Meeting Observation Tool is intended to support agencies in evaluating quality of and adherence to intended practice of child and family team (CFT) meetings. Results can be used to provide information regarding the current status/progress of CFT implementation, guide the work of agency CFT implementation or leadership teams, identify workforce development and organizational support needs, and support Continuous Quality Improvement (CQI) processes. Observers of the CFT will complete throughout the duration of CFT observation.
Knoll and Van Dick Silence Measure | through study completion, ~9 months
  Knoll and Van Dick's 2-Item Silence Measure present scales to assess acquiescent silence and quiescent silence. Participants respond on a scale ranging from 1=strongly disagree to 7=strongly agree, and scale scores are computed by calculating the average item response.

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego - IN STEP Children's Mental Health Research Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sklar M, Kenneally R, Aarons GA, Fettes DL. Applying after-action reviews to child and family teams to improve mental health service linkage within child welfare services: a study protocol. Implement Sci Commun. 2023 Oct 5;4(1):121. doi: 10.1186/s43058-023-00479-3. PMID 37798808